CLINICAL TRIAL: NCT02198313
Title: A Multiple Increasing Dose Safety and Tolerability Study After Inhalation Administration of BIIX 1 XX (100 µg, 200 µg, 400 µg b.i.d. for 14 Days ) in Healthy Male Volunteers (Randomised, Double-blind Within Each Dose Group, Placebo-controlled, Parallel-group)
Brief Title: A Multiple Increasing Dose Safety and Tolerability Study After Inhalation Administration of BIIX 1 XX in Healthy Male Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1150.3
Record Dates: First submitted 2014-07-22; First posted 2014-07-23 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Healthy

ARMS (4):
- BIIX 1 XX - D1 (Experimental)
  Interventions: Drug: BIIX 1 XX - D1
- BIIX 1 XX - D2 (Experimental)
  Interventions: Drug: BIIX 1 XX - D2
- BIIX 1 XX - D3 (Experimental)
  Interventions: Drug: BIIX 1 XX - D3
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIIX 1 XX - D1
  Arms: BIIX 1 XX - D1
Drug: BIIX 1 XX - D2
  Arms: BIIX 1 XX - D2
Drug: BIIX 1 XX - D3
  Arms: BIIX 1 XX - D3
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objective of the present study is to obtain information about the safety and tolerability of multiple increasing doses of BIIX 1 XX and to obtain preliminary pharmacokinetic data

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers who have Broca-Indices within +-20%
* Participants in the age range between 21 to 50 years
* In accordance with Good Clinical Practice (GCP) and local legislation each volunteers are supposed to give their written informed consent prior to admission to the study. Subsequently each subject was to receive a complete medical examination (including blood pressure, pulse rate, medical history, documentation of demographics, inclusion/exclusion criteria and concomitant therapy) as well as a 12-lead Electrocardiogram (ECG)
* Haematopoietic, hepatic and renal function test will be carried out in the laboratory
* The subjects will fast for 12 hours before collection of specimens for all laboratory evaluations. The above mentioned examinations will be performed within 14 days before the first administration of the test substance

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate or ECG) or laboratory tests deviating form normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of a drug with a long half-life (>= 24 hours) within at least one month or less than ten half-lives of the respective drug before enrolment in the study
* Use of any drugs which might influence the results of the trial within seven days prior to administration or during the trial
* Participation in another trial with an investigational drug within the last two months prior to the start of the study
* Smoker (> 10 cigarettes or 3 cigars or 3 pipes/day)
* Inability to refrain from smoking on study days
* History of alcohol abuse and/or alcohol abuse
* Drug abuse
* Blood donation (>100 ml) within four weeks prior to administration
* Other disease or abnormality of clinical relevance
* Excessive physical activities within two weeks prior to administration or during the trial

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 1999-04; Primary Completion 1999-04 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | up to day 28
Number of subjects with abnormal changes in laboratory parameters | up to day 21
Number of subjects with clinically significant changes in vital signs (blood pressure, pulse rate) | up to day 21
Number of subjects with clinically significant changes in ECG (Electrocardiogram) | up to 21 days

SECONDARY OUTCOMES:
AUC (Total Area under the plasma drug concentration time curve) | up to 336 hours after last drug administration
Cmax (maximum observed concentration of the analyte in plasma) | up to 336 hours after last drug administration
tmax (Time from dosing to the maximum concentration of the analyte in plasma) | up to 336 hours after last drug administration
t½ (Terminal half-life of the analyte in plasma) | up to 336 hours after last drug administration
MRT (mean time of residence of drug molecules in the body ) | up to 336 hours after last drug administration
CL (Total clearance of the analyte in plasma following extravascular administration) | up to 336 hours after last drug administration